CLINICAL TRIAL: NCT07235423
Title: Predictors of Post-Thrombectomy Cognitive Impairment in Acute Ischemic Stroke Patients : a Prospective Cohort Study
Brief Title: Predictors of Post-Thrombectomy Cognitive Impairment in Acute Ischemic Stroke Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammad Ahmad Mohammad Korayem, Assistant lecturer, Assiut University
Other Study IDs: CogEVT25
Record Dates: First submitted 2025-09-19; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Stroke, Acute
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postthrombectomy: All patients wgo underwent endovascular thrombectomy under standard care will be assessed for cognitive function at 3 time points

SUMMARY:
This prospective cohort study investigates predictors of post-stroke cognitive impairment (PSCI) in patients undergoing endovascular thrombectomy (EVT) for acute ischemic stroke due to large vessel occlusion. Adult patients with successful reperfusion (mTICI 2b-3) will be followed at 3 and 6 months to assess cognition, functional recovery, and depression. Predictors across clinical, procedural, radiological, and laboratory domains will be analyzed. The study aims to identify risk factors for PSCI, estimate its prevalence, and evaluate its impact on outcomes.

DETAILED DESCRIPTION:
Post-stroke cognitive impairment (PSCI) is a major cause of long-term disability, affecting up to 40% of ischemic stroke survivors. Large vessel occlusion (LVO) strokes, often treated with endovascular thrombectomy (EVT), carry a particularly high risk of cognitive sequelae. While EVT has proven efficacy in improving functional outcomes, its effect on cognitive outcomes remains underexplored.

This prospective observational cohort study will enroll approximately 120 adult patients (≥18 years) with anterior circulation LVO undergoing EVT at Assiut University Hospital. Eligible participants must achieve successful reperfusion (mTICI 2b-3) and provide consent. Patients with severe aphasia, coma, pre-existing dementia, non-ischemic etiologies, or early death (within 72 hours) will be excluded.

Participants will undergo systematic assessment of cognitive function (MoCA-Arabic, Oxford Cognitive Screening if MoCA <26), functional status (mRS, Barthel Index), and mood (HADS-Arabic) at baseline, 3 months, and 6 months. Clinical data (demographics, vascular risk factors, NIHSS, time metrics), procedural details (technique, procedure time, number of passes, anesthesia type, hemodynamic stability, complications), radiological parameters (infarct site and volume, ASPECTS, WMH by Fazekas score, cortical atrophy, microbleeds), and laboratory markers (CRP, ESR, lipid profile, HbA1C, uric acid, D-dimer, CBC) will be collected.

The primary objective is to identify predictors of PSCI at 3-6 months after thrombectomy. Secondary objectives include estimating the prevalence of PSCI in this population and analyzing its association with functional outcomes and depression. Statistical analysis will include univariate and multivariate regression models adjusting for potential confounders such as age, education, and infarct volume.

Ethical approval has been obtained from the Faculty of Medicine, Assiut University Ethics Committee. Written informed consent will be obtained from all participants, and confidentiality will be strictly maintained.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years).
2. Acute ischemic stroke due to anterior circulation LVO confirmed by imaging undergoing EVT per guidelines.
3. Successful reperfusion (mTICI 2b-3)
4. Able to provide consent.

Exclusion Criteria:

1. Severe aphasia/coma interfering with cognitive assessment.
2. Pre-existing dementia ( using Arabic version of the Short Form of the Informant Questionnaire on Cognitive Decline in the Elderly).
3. Non-ischemic etiology.
4. Death within 72 hours.
5. Refusal to participate in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: As described in inclusion/exclusion criteria
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Cognitive impairment after thrombectomy (MoCA) | 3 months (±2 weeks) and 6 months (±2 weeks) post-thrombectomy
  Cognitive status will be assessed using the Arabic version of the Montreal Cognitive Assessment (MoCA, score range 0-30, with scores <26 indicating impairment). The primary outcome will be the prevalence of post-stroke cognitive impairment (PSCI) among thrombectomy patients.

SECONDARY OUTCOMES:
Domain-specific cognitive performance (OCS) | 3 months (±2 weeks) and 6 months (±2 weeks) post-thrombectomy
  For participants scoring <26 on MoCA, the Oxford Cognitive Screen (OCS) will be administered to evaluate specific domains of cognition (attention, executive function, memory, language, visuospatial ability).
Depression and anxiety symptoms (HADS) | 3 months (±2 weeks) and 6 months (±2 weeks) post-thrombectomy
  Psychological status will be measured using the Hospital Anxiety and Depression Scale (HADS, score range 0-21 per subscale). Outcomes will include mean scores and prevalence of clinically significant symptoms.
Functional independence (Barthel Index) | 3 months (±2 weeks) and 6 months (±2 weeks) post-thrombectomy
  Functional status will be assessed using the Barthel Index (score range 0-100). Higher scores indicate greater independence in activities of daily living.
Global disability (modified Rankin Scale) | 3 months (±2 weeks) and 6 months (±2 weeks) post-thrombectomy
  Global disability will be measured using the modified Rankin Scale (mRS, score range 0-6, with 0 indicating no symptoms and 6 indicating death).
Infarct volume (DWI MRI) | Within 24-72 hours post-thrombectomy
  Infarct size will be quantified using diffusion-weighted MRI, measured in milliliters.
White matter hyperintensity (Fazekas score) | Within 24-72 hours post-thrombectomy
  White matter disease burden will be assessed using the Fazekas score (0-3 scale) on FLAIR MRI
CRP | Within 24-72 hours post-thrombectomy
  C-reactive protein (CRP, mg/L)
Lipid profile | Within 24-72 hours post-thrombectomy
  lipid profile (mg/dL)
Ddimer | Within 24-72 hours post-thrombectomy
  D-dimer (µg/mL)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://doi.org/10.3389/fnagi.2024.1359792
- See also: Related Info — http://doi.org/10.1016/j.ahr.2025.100232
- See also: Related Info — https://doi.org/10.1186/s12883-021-02117-8
- See also: Related Info — https://doi.org/10.20471/acc.2023.62.s1.05
- See also: Related Info — https://doi.org/10.1017/S1041610204000390